CLINICAL TRIAL: NCT07088159
Title: Intermediate-size Patient Population Expanded Access Protocol for SPG302 in Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Intermediate-size Patient Population Expanded Access Protocol
Status: Available | Type: Expanded Access
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Other Study IDs: SPG302-ALS-ISEAP
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Expanded Access Protocol; synapse; ALS (Amyotrophic Lateral Sclerosis); neural connectivity
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: SPG302 — 300 mg SPG302 will taken by mouth once daily.

SUMMARY:
The purpose of this Expanded Access Program is to provide SPG302 to ALS patients who are not eligible to enroll in an ALS clinical trial. This Expanded Access Program will assess safety and tolerability, and clinical efficacy of SPG302.

DETAILED DESCRIPTION:
This is a multi-site, intermediate-size patient population expanded access protocol developed to provide compassionate use access to SPG302 to adult patients with ALS who have progressed following available standard of care.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosis
* Age 18 -80 years at time of signing informed consent form
* Ineligible for other interventional ALS clinical research participation
* Vital Capacity less than 50% of predicted capacity for age, height, and sex
* If currently taking standard of care treatment for ALS, must be on stable dose for at least 30 days prior to taking SPG302.
* Life expectancy of at least 6 months, according to Investigator's judgement

Exclusion Criteria:

* Clinically significant and/or unstable medical condition (other than ALS) that would pose a risk to the patient
* Known ongoing or clinically uncontrolled cardiac disease
* Clinically significant liver disease
* Clinical significant cognitive impairment or neurological disorder, as determined by Investigator judgement
* Concomitant use of another investigational medical product for treatment of ALS
* Unable to reliably and regularly swallow whole oral medications on a daily basis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Mayo Scottsdale, Scottsdale, Arizona
  - Cedar-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Nova Southeastern University, Davie, Florida
  - Synapticure, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Health, Summit, New Jersey
  - Columbia University Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - VCU ALS Research Group, Henrico, Virginia